CLINICAL TRIAL: NCT03193437
Title: A Phase 2, Open-label Study of Selinexor (KPT-330) in Patients With Advanced Thymic Epithelial Tumor (TET) Progressing After Primary Chemotherapy (SELECT)
Brief Title: Selinexor in Patients With Advanced Thymic Epithelial Tumor Progressing After Primary Chemotherapy
Acronym: SELECT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Georgetown University (Other)
Collaborators: Hackensack Meridian Health (Other); Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0622
Record Dates: First submitted 2017-06-19; First posted 2017-06-20 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-04

CONDITIONS: Thymoma; Advanced Thymic Epithelial Tumor
Keywords: Thymus; Selinexor; KPT-330
MeSH Terms: conditions — Thymoma | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selinexor (Experimental): Open Label Selinexor 40 mg
  Interventions: Drug: Open Label Selinexor

INTERVENTIONS:
Drug: Open Label Selinexor — Selinexor 40 mg oral tablets will be administered twice weekly, either on Monday/Wednesday, Tuesday/Thursday, Wednesday/Friday, Thursday/Saturday, or Friday/Sunday in a 3-weeks-on and 1-week-off schedule.
  Other Names: KPT-330

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and effectiveness of selinexor in patients with advanced thymic epithelial tumor progressing after primary chemotherapy. This is a multicenter, open label phase II trial that uses a Simons two stage design. The study population is adults with histologically confirmed, advanced, inoperable TETs who are progressing after treatment with at least one platinum containing chemotherapy regimen.

This study is comprised of 2 similar phase II trials, one running in US (25 patients) and one running in EU (25 patients):

There are two study arms:

Arm A: Thymoma

* Stage 1: 15 patients
* Stage 2: 10 patients

Arm B: Thymic carcinoma

* Stage 1: 15 patients
* Stage 2: 10 patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced TET (thymoma)
* Progression after Primary Chemotherapy
* No more than two previous lines (Neoadjuvant or chemoradiotherapy will count as one line if disease progression has occurred within 6 months)
* Inoperable per local Investigator (Masaoka Stage III or IV)
* Progression after treatment with least one platinum containing chemotherapy regimen
* Measurable disease (RECIST 1.1)
* Age ≥18 years
* ECOG PS <2
* Patients must have recovered from the toxic effects of prior therapy at the time of initiation of the study drug unless toxicity is stable.
* A 4 weeks or five half lives interval from any investigational agents or cytotoxic chemotherapy to start of study is required
* Signed informed consent
* Adequate bone marrow function and organ function:

  * Hematopoietic function: total white blood cell count (WBC) ≥ 3000/mm³, absolute neutrophil count (ANC) ≥ 1500/mm³, platelet count ≥ 100,000/mm²; Hemoglobin > 9.0 gm/dL
  * Hepatic function: bilirubin < 1.5 times the upper limit of normal (ULN), ALT < 2.5 times ULN or ALT < 5.0 times ULN in the presence of liver metastases
  * Creatinine clearance > 30 ml/min according to Cockcroft-Gault
* Patients of childbearing potential must agree to use adequate birth control during and for 7 months after participation in this study

Exclusion Criteria:

* No significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy, including

  * Unstable cardiovascular function
  * Known active hepatitis A, B, or C infection; or known to be positive for HCV RNA or HBsAg (HBV surface antigen)
  * Markedly decreased visual acuity
  * Active infection requiring intravenous antibiotics
* Pregnancy or breast-feeding
* Symptomatic brain metastasis requiring corticosteroids
* Uncontrolled autoimmune disorders. Patients with autoimmune disorders under control on medication may be included. Patients with pure red cell aplasia may be included if haemoglobin levels are relatively stable on transfusions or medication
* Significantly diseased or obstructed gastrointestinal tract, malabsorption, uncontrolled vomiting or diarrhea or inability to swallow oral medications
* No dehydration of NCI-CTCAE grade ≥ 1
* Serious psychiatric or medical conditions that could interfere with treatment.
* No history of organ allograft
* No concurrent therapy with approved or investigational anticancer therapeutics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chul Kim, MD, Study Chair — Georgetown University
Locations (2):
- United States (2):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center - Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Selinexor
Started | 8
Completed | 0
Not Completed | 8
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 2
Not completed — Disease Progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Selinexor
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To determine the overall response rate per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR+ PR.
Time Frame: 24 months
Measure: Number; unit: percentage of patients
Arm/Group | Selinexor
Number analyzed (Participants) | 8
percentage of patients | 0

2. Secondary Outcome: Overall Response Rate
Description: To determine the overall response rate to according to modified ITMIG response criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT and MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 24 months
Measure: Number; unit: percent of participants
Arm/Group | Selinexor
Number analyzed (Participants) | 8
percent of participants | 0

3. Secondary Outcome: 6 Month Progression Free Survival Rate
Description: To determine six months progression free survival of patients with TET treated with selinexor
Time Frame: 6 months
Measure: Number; unit: percent
Arm/Group | Selinexor
Number analyzed (Participants) | 8
percent | 55.6

4. Secondary Outcome: 24 Month Overall Survival Rate
Description: To determine overall survival of patients with TET treated with selinexor
Time Frame: 24 months
Measure: Number; unit: percent
Arm/Group | Selinexor
Number analyzed (Participants) | 8
percent | 57.1

5. Secondary Outcome: Adverse Events
Description: The number of adverse events as determined by Common Terminology Criteria for Adverse Events (CTCAEs) version 4.03
Time Frame: 24 months
Measure: Number; unit: Adverse events
Arm/Group | Selinexor
Number analyzed (Participants) | 8
Adverse events | 93

ADVERSE EVENTS:
Time Frame: From the time of consent to 30 days following the last dose of study treatment (max 24 months).
Arm/Group | Selinexor
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 5/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selinexor (N=8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 2 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selinexor (N=8)
Anemia (Blood and lymphatic system disorders) | 4 (10)
Cardiac Disorders other, specify (Cardiac disorders) | 1 (1) — QTc Prolongation
Cataract (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — light sensitivity
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 7 (10)
Vomiting (Gastrointestinal disorders) | 3 (3)
asthenia (General disorders) | 1 (2)
lightheadedness (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — sore throat, productive cough
Mucosal infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 3 (3)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Tardive dyskinesia
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT03193437/Prot_SAP_000.pdf